CLINICAL TRIAL: NCT01134081
Title: Expression of Angiogenic Biomarkers During Healing of Intra-Oral Soft Tissue Engineered Grafts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Organogenesis (Industry)
Responsible Party: Principal Investigator, William Giannobile, Chair, Department of Periodontics & Oral Medicine Najjar Endowed Professor of Dentistry and Biomedical Engineering, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 06-PER-002-CTX Bio Adjunct
Record Dates: First submitted 2010-05-20; First posted 2010-05-31 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2017-08-21 (Actual); Status verified 2017-06

CONDITIONS: Gingival Recession
Keywords: gum; recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CelTx™ (Experimental): Living bilayered cell therapy product
  Interventions: Biological: CelTx™
- Free Gingival Grafts (Active Comparator): Harvested tissue from palate
  Interventions: Procedure: Free Gingival Graft

INTERVENTIONS:
Biological: CelTx™ — CelTx™ is a living bilayered cell therapy product. CelTx™ is constructed of Type I bovine collagen (extracted from bovine tendons and subsequently purified) and viable allogeneic human fibroblasts and keratinocytes isolated from human neonatal foreskin. This is applied once in the oral cavity.
  Arms: CelTx™
Procedure: Free Gingival Graft — Harvested tissue from palate
  Arms: Free Gingival Grafts

SUMMARY:
The purpose of this observational research study is to understand more about wound healing of gum tissue. This study was the biomarker study of a small cohort of study participants derived from NCT01547962 (completed). Two surgical sites of each patient were randomly selected to receive CelTx™ as a donor material in one site and conventional autograft using keratinized tissue from the palate as the donor material at the contralateral (opposite side) site. Fluids collected from between a tooth and the gum and directly from wounds contain proteins that occur in different levels as the wound healing process proceeds. In this research study wound fluid will be collected from the donor palate site (roof of your mouth) and the treated sites on your gum before and after placement of CelTx and conventional treatment (tissue from the roof of your mouth) to measure which proteins and how much of each are present during the first 4 weeks of wound healing.

DETAILED DESCRIPTION:
In a clinical trial designed to evaluate the safety and effectiveness of rhPDGF-BB to promote soft and hard tissue engineering of the periodontium, the subjects provided gingival crevicular fluid (GCF) or periodontal wound fluid (WF) and the results demonstrated contrasting inducible expression patterns of PDGF-AB, VEGF, and ICTP during periodontal healing [17, 24, 25]. However, little is known regarding the release of these molecules into local periodontal wound fluid during tissue-engineered grafts.

The aim of this study is to determine the presence and influence of angiogenic biomarkers, such as PDGF, VEGF, and FGF, involved in the wound healing process of tissue engineered grafts in the treatment of subjects (with recession-type defects) who have an insufficient zone of attached gingival associated with at least two nonadjacent teeth.

STUDY OBJECTIVES The purpose of this pilot study is to compare the expression of angiogenic biomarkers involved in the wound healing process of 2 different periodontal surgical approaches: 1) CelTx™ (living bilayered cell therapy product) and 2) free gingival grafts

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed informed consent to participate in Organogenesis Clinical Protocol 06-PER-002-CTX.
* Subject has signed informed consent to participate in this adjunct bio-marker study.
* Subject is willing to comply with the additional study visits at weeks 2 and 3 as required by this study.

Exclusion Criteria:

- Subject requires antibiotic prophylaxis for routine dental procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Neiva, DDS, MS, Principal Investigator — University of Michigan
Locations (1):
- Michigan Center for Oral Health Research, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Morelli T, Neiva R, Nevins ML, McGuire MK, Scheyer ET, Oh TJ, Braun TM, Nor JE, Bates D, Giannobile WV. Angiogenic biomarkers and healing of living cellular constructs. J Dent Res. 2011 Apr;90(4):456-62. doi: 10.1177/0022034510389334. Epub 2011 Jan 19. PMID 21248359

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 subjects were enrolled. All 44 subjects participated in both arms/groups for a total of 88 surgical sites. 2 surgical sites of each patient were randomly selected to receive LCC as a donor material in 1 site and a conventional autograft using keratinized tissue from the palate as the donor material at the contralateral site.
Groups:
- CelTx™ & Free Gingival Grafts: CelTx™: Living bilayered cell therapy product Free Gingival Grafts: Harvested tissue from palate
Period: Overall Study
Arm/Group | CelTx™ & Free Gingival Grafts
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Units Other Than Participants: Surgical sites
Arm/Group | CelTx™ & Free Gingival Grafts
Number analyzed (Participants) | 44
Number analyzed (Surgical sites) | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 25
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Differences in Angiogenic Biomarkers
Description: Within-subject difference between the concentrations at the CelTX and Free Gingival Graft areas
Time Frame: 5 time-points: pre-surgical, week(s) 1, 2, 3 and 4
Population: 44 subjects were enrolled. All 44 subjects participated in both arms/groups for a total of 88 surgical sites. 2 surgical sites of each patient were randomly selected to receive LCC as a donor material in 1 site and a conventional autograft using keratinized tissue from the palate as the donor material at the contralateral site.
Measure: Mean (Standard Error); unit: ng/mL
Units Other Than Participants: Surgical sites
Arm/Group | CelTx™ | Free Gingival Grafts
Number analyzed (Participants) | 44 | 44
Number analyzed (Surgical sites) | 44 | 44
ng/mL
  VEGF-pre-surgical | 0.51 (.07) | .69 (.15)
  VGEF-week 1 | 1.04 (.24) | .67 (.12)
  VGEF-week 2 | .28 (.06) | .16 (.04)
  VGEF-week 3 | .14 (.03) | .11 (.03)
  VGEF-week 4 | .1 (.02) | .06 (.02)
  Angiogenin (ANG)-pre-surgical | 6.19 (.97) | 5.60 (.82)
  Angiogenin (ANG)-week 1 | 8.32 (1.26) | 7.09 (1.24)
  Angiogenin (ANG)-week 2 | 3.67 (.65) | 2.56 (.54)
  Angiogenin (ANG)-week 3 | 1.92 (.30) | 1.85 (.36)
  Angiogenin (ANG)-week 4 | 1.34 (.23) | 1.58 (.38)
  IL-8-pre-surgical | 1.29 (.21) | 1.31 (.22)
  IL-8-week 1 | 5.6 (.76) | 4.44 (.72)
  IL-8-week 2 | .58 (.15) | .31 (.09)
  IL-8-week 3 | .19 (.07) | .15 (.06)
  IL-8-week 4 | .11 (.03) | .11 (.04)
  FGF-2-pre-surgical | .65 (.12) | .72 (.17)
  FGF-2-week 1 | 1.36 (.51) | .85 (.17)
  FGF-2-week 2 | .4 (.11) | .34 (.11)
  FGF-2-week 3 | .20 (.06) | .29 (.08)
  FGF-2-week 4 | .18 (.07) | .24 (.08)
  Angiostatin (ANT)-pre-surgical | 6728.08 (1996.62) | 7931.32 (2813.77)
  Angiostatin (ANT)-week 1 | 12330.29 (3523.17) | 3871.60 (782.5)
  Angiostatin (ANT)-week 2 | 3059.87 (1037.32) | 1524.59 (654.12)
  Angiostatin (ANT)-week 3 | 1668.22 (605.07) | 1682.54 (453.33)
  Angiostatin (ANT)-week 4 | 1527.26 (507.75) | 1183.51 (441.75)
  TIMP-1-pre-surgical | 9.14 (1.09) | 8.56 (1.25)
  TIMP-1-week 1 | 16.63 (1.68) | 14.68 (1.77)
  TIMP-1-week 2 | 7.81 (1.42) | 5.60 (.93)
  TIMP-1-week 3 | 4.63 (.94) | 3.98 (.77)
  TIMP-1-week 4 | 3.98 (.72) | 3.58 (.73)
  TIMP-2-pre-surgical | 6.85 (1.51) | 11.11 (4.18)
  TIMP-2-week 1 | 17.13 (3.47) | 9.91 (2.14)
  TIMP-2-week 2 | 3.70 (.95) | 2.41 (.77)
  TIMP-2-week 3 | 2.16 (.70) | 1.43 (.46)
  TIMP-2-week 4 | 1.50 (.52) | .93 (.34)
  GM-CSF-pre-surgical | 59.48 (19.53) | 50.27 (13.97)
  GM-CSF-week 1 | 99.85 (21.57) | 102.02 (24.65)
  GM-CSF-week 2 | 93.20 (21.38) | 93.81 (20.36)
  GM-CSF-week 3 | 91.16 (20.76) | 86.16 (18.34)
  GM-CSF-week 4 | 71.81 (16.76) | 80.34 (16.12)
  IP-10-pre-surgical | .78 (.36) | .21 (.07)
  IP-10-week 1 | .03 (.02) | .5 (.45)
  IP-10-week 2 | .39 (.29) | .08 (.08)
  IP-10-week 3 | .18 (.12) | .02 (.01)
  IP-10-week 4 | .01 (.01) | .01 (.01)

2. Primary Outcome: Differences in Angiogenic Biomarkers: PDGF-BB
Description: Within-subject difference between the concentrations at the CelTX and Free Gingival Graft areas
Time Frame: 5 time-points: pre-surgical, week(s) 1, 2, 3 and 4
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | CelTx™ | Free Gingival Grafts
Number analyzed (Participants) | 44 | 44
pg/mL
  Pre-surgical | 10.59 (3.06) | 9.73 (3.41)
  Week 1 | 51.82 (20.41) | 28.92 (13.73)
  Week 2 | 4.50 (3.03) | 2.33 (1.00)
  Week 3 | 2.15 (.83) | 1.01 (.44)
  Week 4 | .86 (.43) | .87 (.50)

ADVERSE EVENTS:
Time Frame: 6 months
Description: No adverse or serious adverse events were observed.
Arm/Group | CelTx™ | Free Gingival Graft
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/44

LIMITATIONS AND CAVEATS:
Although the present study compared the differences in angiogenic biomarker expression between LCC and autograft, it is important to understand that both LCC and autograft heal by two different healing processes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes